CLINICAL TRIAL: NCT06962059
Title: Vaginal Metabolome Healthy Volunteers Study
Brief Title: Healthy Volunteers Study
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 01025
Record Dates: First submitted 2025-04-10; First posted 2025-05-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer; Genetic Predisposition to Disease
Keywords: vaginal metabolome; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteer: Females 30 or older who do not have a genetic predisposition to ovarian cancer, are unaffected by cancer, and have not had bilateral oophorectomy.
  Interventions: Other: Self-Administered Sample Collection

INTERVENTIONS:
Other: Self-Administered Sample Collection — Participants will collect vaginal swabs and a stool sample.

SUMMARY:
The purpose of this study is to examine the role of the bacterial environments and metabolites in the early detection and prediction of ovarian cancer development. Vaginal swabs and stool samples will be collected from healthy volunteers, or those without a known ovarian cancer diagnosis or genetic ovarian cancer risk. These samples will be compared to samples from participants with increased cancer risk and ovarian cancer diagnoses.

DETAILED DESCRIPTION:
This study will examine the role of the microbiome and its metabolites in early detection and prediction of ovarian cancer development. It has been previously shown that the composition and function of the microbiome may play a role in the development and progression of several types of cancer. One proposed mechanism by which the microbiome may contribute to cancer development is through the production of certain metabolic byproducts. Such metabolites produced or modified by the microbiome have emerged as a prominent factor with potential local and systemic effects on the host, and were proposed to mediate the microbiome's contribution to cancer development. Microbial metabolites can promote cancer development by activating signaling pathways that promote cell growth and survival. In addition, the microbiota affects carcinogenesis through the release of carcinogenic molecules, such as genotoxins, and through the production of tumor-promoting metabolites. Furthermore, microbial metabolites have been studied as potential biomarkers for cancer, with some research suggesting that certain microbial metabolites may be able to distinguish between healthy individuals and those with cancer. The microbiome of the female reproductive tract is relatively understudied compared to the gut microbiome, but recent studies have shown that it is present and diverse in various parts of the reproductive tract such as the vagina, cervix, and fallopian tubes. however, a microbiome or metabolome signature predictive of ovarian cancer has not yet been established. Eligible individuals will be consented to provide a one-time, self-administered vaginal swab sample and stool sample. Clinical research assistants/coordinators, genetic counselors, and/or study physicians will consent patients and process and store the samples of consented participants. Participants will be provided a stool collection kit at the time of consent with instructions for providing the sample and sending it back to the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* has ovaries

Exclusion Criteria:

* genetic mutations which increase risk of ovarian cancer: BRCA1/2, BRIP1, PALB2, Lynch Syndrome (MLH1, MSH2/EPCAM, MSH6) and ATM
* no genetic testing results or unknown genetic status
* prior cancer diagnosis
* prior cancer treatment
* HRT use
* Antibiotic use (1 month prior to providing sample)

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eligible participants will be patients of the Cancer Risk Evaluation Program at the Abramson Cancer Center. Patients who meet the above criteria will be approached to participate as healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Microbiome Involvement | One-time sample donation of vaginal swabs collected at the time of the patient's appointment. A subsequent stool sample will be provided within a week of the vaginal swab.
  Investigate the involvement of the microbiome and associated metabolites in ovarian cancer.
Predictive Model | One-time sample donation of vaginal swabs collected at the time of the patient's appointment. A subsequent stool sample will be provided within a week of the vaginal swab.
  Generate a predictive model for ovarian cancer risk and progression. Healthy volunteers will provide a control group to compare to BRCA-carrier and affected cohorts consented through the CREP Biobank study in order to mechanistically understand the function of the identified metabolites in disease prevention, initiation, progression, and treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Domchek, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data of patients samples, survey answers, and complementary medical information will be shared with investigators at Stanford and Columbia. This information will be used to identify factors for analysis such as prescribed medications, treatment types and timeframes, among others.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared with investigators three months after enrollment is complete. This should provide time for enrolled subjects to complete participation, ensure all data entry is complete, and that all data from records is obtained.

REFERENCES:
- [Background] Manasa G, Mascarenhas RJ, Shetti NP, Malode SJ, Aminabhavi TM. Biomarkers for Early Diagnosis of Ovarian Carcinoma. ACS Biomater Sci Eng. 2022 Jul 11;8(7):2726-2746. doi: 10.1021/acsbiomaterials.2c00390. Epub 2022 Jun 28. PMID 35762531
- [Background] Manganaro L, Celli V, Viggiani V, Berardelli E, Granato T, Tartaglione S, Farina A, Catalano C, Angeloni A, Anastasi E. CT imaging phenotypes linked to CA125 and HE4 biomarkers are highly predictive in discriminating between hereditary and sporadic ovarian cancer patients. Tumour Biol. 2022;44(1):171-185. doi: 10.3233/TUB-211557. PMID 36093649
- [Background] Menon U, Karpinskyj C, Gentry-Maharaj A. Ovarian Cancer Prevention and Screening. Obstet Gynecol. 2018 May;131(5):909-927. doi: 10.1097/AOG.0000000000002580. PMID 29630008
- [Background] Cullin N, Azevedo Antunes C, Straussman R, Stein-Thoeringer CK, Elinav E. Microbiome and cancer. Cancer Cell. 2021 Oct 11;39(10):1317-1341. doi: 10.1016/j.ccell.2021.08.006. Epub 2021 Sep 9. PMID 34506740
- [Background] Levy M, Thaiss CA, Elinav E. Metabolites: messengers between the microbiota and the immune system. Genes Dev. 2016 Jul 15;30(14):1589-97. doi: 10.1101/gad.284091.116. PMID 27474437
- [Background] Cao Y, Oh J, Xue M, Huh WJ, Wang J, Gonzalez-Hernandez JA, Rice TA, Martin AL, Song D, Crawford JM, Herzon SB, Palm NW. Commensal microbiota from patients with inflammatory bowel disease produce genotoxic metabolites. Science. 2022 Oct 28;378(6618):eabm3233. doi: 10.1126/science.abm3233. Epub 2022 Oct 28. PMID 36302024
- [Background] Kroemer G, McQuade JL, Merad M, Andre F, Zitvogel L. Bodywide ecological interventions on cancer. Nat Med. 2023 Jan;29(1):59-74. doi: 10.1038/s41591-022-02193-4. Epub 2023 Jan 19. PMID 36658422
- [Background] Dmitrieva-Posocco O, Wong AC, Lundgren P, Golos AM, Descamps HC, Dohnalova L, Cramer Z, Tian Y, Yueh B, Eskiocak O, Egervari G, Lan Y, Liu J, Fan J, Kim J, Madhu B, Schneider KM, Khoziainova S, Andreeva N, Wang Q, Li N, Furth EE, Bailis W, Kelsen JR, Hamilton KE, Kaestner KH, Berger SL, Epstein JA, Jain R, Li M, Beyaz S, Lengner CJ, Katona BW, Grivennikov SI, Thaiss CA, Levy M. beta-Hydroxybutyrate suppresses colorectal cancer. Nature. 2022 May;605(7908):160-165. doi: 10.1038/s41586-022-04649-6. Epub 2022 Apr 27. PMID 35477756
- [Background] France M, Alizadeh M, Brown S, Ma B, Ravel J. Towards a deeper understanding of the vaginal microbiota. Nat Microbiol. 2022 Mar;7(3):367-378. doi: 10.1038/s41564-022-01083-2. Epub 2022 Mar 4. PMID 35246662
- [Background] Wang J, Li Z, Ma X, Du L, Jia Z, Cui X, Yu L, Yang J, Xiao L, Zhang B, Fan H, Zhao F. Translocation of vaginal microbiota is involved in impairment and protection of uterine health. Nat Commun. 2021 Jul 7;12(1):4191. doi: 10.1038/s41467-021-24516-8. PMID 34234149
- [Background] Kindschuh WF, Baldini F, Liu MC, Liao J, Meydan Y, Lee HH, Heinken A, Thiele I, Thaiss CA, Levy M, Korem T. Preterm birth is associated with xenobiotics and predicted by the vaginal metabolome. Nat Microbiol. 2023 Feb;8(2):246-259. doi: 10.1038/s41564-022-01293-8. Epub 2023 Jan 12. PMID 36635575
- [Background] Asangba AE, Chen J, Goergen KM, Larson MC, Oberg AL, Casarin J, Multinu F, Kaufmann SH, Mariani A, Chia N, Walther-Antonio MRS. Diagnostic and prognostic potential of the microbiome in ovarian cancer treatment response. Sci Rep. 2023 Jan 13;13(1):730. doi: 10.1038/s41598-023-27555-x. PMID 36639731
- [Background] Zhou B, Sun C, Huang J, Xia M, Guo E, Li N, Lu H, Shan W, Wu Y, Li Y, Xu X, Weng D, Meng L, Hu J, Gao Q, Ma D, Chen G. The biodiversity Composition of Microbiome in Ovarian Carcinoma Patients. Sci Rep. 2019 Feb 8;9(1):1691. doi: 10.1038/s41598-018-38031-2. PMID 30737418
- [Background] Cheng H, Wang Z, Cui L, Wen Y, Chen X, Gong F, Yi H. Opportunities and Challenges of the Human Microbiome in Ovarian Cancer. Front Oncol. 2020 Feb 18;10:163. doi: 10.3389/fonc.2020.00163. eCollection 2020. PMID 32133297
- [Background] Nene NR, Reisel D, Leimbach A, Franchi D, Jones A, Evans I, Knapp S, Ryan A, Ghazali S, Timms JF, Paprotka T, Bjorge L, Zikan M, Cibula D, Colombo N, Widschwendter M. Association between the cervicovaginal microbiome, BRCA1 mutation status, and risk of ovarian cancer: a case-control study. Lancet Oncol. 2019 Aug;20(8):1171-1182. doi: 10.1016/S1470-2045(19)30340-7. Epub 2019 Jul 9. PMID 31300207